CLINICAL TRIAL: NCT00368979
Title: Clinical Evaluation of Dutasteride in Benign Prostatic Hyperplasia: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Comparative Study of GI198745 (Dutasteride) in Subjects With Benign Prostatic Hyperplasia.
Brief Title: Dutasteride (GI198745) In Benign Prostatic Hyperplasia Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI105326
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2009-04-02 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia BPH dutasteride
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dutasteride (Active Comparator)
  Interventions: Drug: Dutasteride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — once daily
  Arms: Dutasteride
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of GI198745 0.5mg given once daily for 52 weeks to Benign Prostatic Hyperplasia (BPH) patients.

ELIGIBILITY:
Inclusion Criteria:

Only subjects who meet all the following criteria during the screening phase will be enrolled in the study.

1. Diagnosis: BPH
2. Age: ≥50 years
3. Gender: Male
4. Estimated prostate volume ≥30cc (by TRUS)
5. I-PSS Symptom Score (total of 7 items) ≥8 points
6. Maximum flow rate (Qmax) ≤15mL/sec (voided volume measured simultaneously ≤150mL)*[1]
7. Patients who meet either of the following regarding tamsulosin HCl use:

   Patients with tamsulosin HCl use:

   Patients who have received tamsulosin HCl continuously for at least 4 weeks and who are likely to continue to take tamsulosin HCl without any change to the dosage and administration of the drug until the end of study treatment.

   Patients without tamsulosin HCl use:

   Patients who haven't received tamsulosin HCl in the past 4 weeks and who are unlikely to use tamsulosin HCl until the end of study treatment.
8. Outpatients
9. Patients who in person have given written consent

Exclusion Criteria:

Patients who apply to any of the following criteria during the screening phase will not be enrolled in the study.

1. Post void residual volume >250mL (by suprapubic ultrasound).
2. History of AUR within the previous 12 weeks.
3. Evidence or history of prostate cancer.
4. PSA >10ng/mL [in patients with PSA >4ng/mL, the presence of prostate cancer should be ruled out by the investigator/subinvestigator. DRE and free/total PSA ratio should be considered, and prostate biopsy be conducted if necessary].
5. Previous surgery (including balloon dilatation, thermotherapy and stent placement) or minimally invasive techniques for BPH.
6. Any causes other than BPH, which may in the judgment of the investigator/subinvestigator, affect evaluation of symptoms or urine flow (e.g., neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute/chronic prostatitis, acute/chronic urinary tract infection).
7. History of any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias*[2], congestive heart failure or cerebrovascular accident within the previous 6 months; or diabetes mellitus or peptic ulcer uncontrollable with medical treatment.
8. Liver function tests (AST, ALT, AL-P) >2 times the upper limit of normal.
9. Serum cleatinine >1.8mg/dL.
10. Use of any antiandrogen (e.g., chlormadinone acetate, allylesterenol) for BPH within the previous 12 months.
11. Use of a1-adrenoceptor blockers excluding tamsulosin HCl (e.g., prazosin HCl, urapidil slow-release capsule formulation, terazosin HCl, naftopidil), plant extract preparations for treatment of BPH (e.g., Eviprostat, cernitin pollen extract), herbal medicines (e.g., hachimi-jio-gan, gosha-jinki-gan), other drugs (e.g., Paraprost), and dietary or herbal supplements (e.g., saw palmetto) for relief of BPH symptoms within the previous 4 weeks.

Use of a-adrenoceptor agonists (e.g., pseudoephedrine, phenyle

* [1] Subjects with voided volume <150 mL at Qmax measurement cannot be enrolled in the study and may undergo re-measurement of Qmax before the visit for Week 0 for study entry.
* [2] Of "Degree II" according to "Grading of Side Effects (PMSB Notification No. 80 dated June 29, 1992) or equivalent (Appendix 4).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2006-02-17; Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Japan (8):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Background] Tsukamoto T, Endo Y, Narita M. Efficacy and safety of dutasteride in Japanese men with benign prostatic hyperplasia. Int J Urol. 2009 Sep;16(9):745-50. doi: 10.1111/j.1442-2042.2009.02357.x. Epub 2009 Aug 5. PMID 19674165

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects who took no study medication capsule once daily for 52 weeks followed by up to 16 weeks of post-dosing assessments.
- Dutasteride: Subjects who took dutasteride, study medication of 0.5 mg capsule once daily for 52 weeks followed by up to 16 weeks of post-dosing assessments.
Period: Overall Study
Arm/Group | Placebo | Dutasteride
Started | 185 | 193
Completed | 160 | 163
Not Completed | 25 | 30
Not completed — Adverse Event | 9 | 16
Not completed — Lack of Efficacy | 5 | 3
Not completed — Other | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dutasteride | Total
Number analyzed (Participants) | 181 | 184 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (6.76) | 68.0 (6.07) | 67.4 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 181 | 184 | 365
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese | 181 | 184 | 365

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) at Week 52
Description: The International Prostate Symptom Score (I-PSS) consists of 7 verified questions concerning urinary symptoms and one quality of life question scored from 0 to 5(0=Not at All, to 5=Almost Always). The total score can range from 0 to 35. Score of 1-7=Mild, 8-19=Moderate, 20-35=Severe.
Time Frame: Baseline and Week 52
Population: The Full Analysis Set (FAS) which consisted of all randomized participants with a history excluding those who received no dose of the investigational product and who had no baseline or post baseline IPSS data. Last Observation Carried Forward (LOCF) method for lost data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 181 | 184
score on a scale | -3.6 (5.72) | -5.5 (5.94)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Net) = -1.6, 95% CI [-2.7 to -0.5]

2. Secondary Outcome: Percent Change From Baseline in Prostate Volume at Week 52
Description: Prostate volume measurements by transrectal ultrasound (TRUS). Average prostate volume (55cc). The Ultrasound scans the prostate in the transverse plane while moving in the cephalocaudal direction of the prostate. The height and width of the prostate section with the greatest surface area is recorded.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeters (cc)
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 180 | 183
cubic centimeters (cc) | -8.9 (18.76) | -31.5 (16.85)

3. Secondary Outcome: Number of Participants With IPSS Improvement From Baseline at Week 52
Description: Improvement is defined as greater than or equal to a 2 point increase in participants total score on the I-PSS questionaire.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 181 | 184
participants
  Improvement >=2 Points | 113 | 139
  Improvement >=3 Points | 102 | 128
  Improvement >=4 Points | 82 | 115
  Improvement >=5 Points | 75 | 94
  Improvement >=6 Points | 62 | 82
  Improvement >=20% | 99 | 122
  Improvement >=25% | 84 | 114
  Improvement >=30% | 71 | 106
  Improvement >=40% | 54 | 86
  Improvement >=50% | 39 | 67
  Improvement >=75% | 7 | 17

4. Secondary Outcome: Change From Baseline in Maximum Urine Flow Rate (Qmax) at Week 52
Description: Maximum Urine Flow Rate (Qmax) is the peak flow in milliliters per second.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters per second (mL/sec)
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 181 | 184
milliliters per second (mL/sec) | 0.6 (3.82) | 2.2 (4.89)

5. Secondary Outcome: Number of Participants With Qmax Improvement From Baseline at Week 52
Description: Improvement was defined as an increase in Qmax by greater than or equal to 1 mL/sec
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 179 | 183
participants
  Improvement >=1 mL/sec | 79 | 103
  Improvement >=2 mL/sec | 56 | 86
  Improvement >=2.5 mL/sec | 45 | 73
  Improvement >=3 mL/sec | 44 | 70
  Improvement >=4 mL/sec | 29 | 53
  Improvement >=5 mL/sec | 22 | 44
  Improvement >=10 mL/sec | 4 | 11
  Improvement >=30% | 41 | 63

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in all participants who received at least one dose of the investigational product.
Arm/Group | Placebo | Dutasteride
Serious Adverse Events (participants affected / at risk) | 8/184 | 20/193
Other Adverse Events (participants affected / at risk) | 116/184 | 124/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | Dutasteride (N=193)
Colonic polyp (Gastrointestinal disorders) | 0 | 3
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Microscopic polyangiitis (Vascular disorders) | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=184) | Dutasteride (N=193)
Nasopharyngitis (Infections and infestations) | 78 | 80
Diarrhoea (Gastrointestinal disorders) | 16 | 19
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 14 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 12
Constipation (Gastrointestinal disorders) | 12 | 13
Eczema (Skin and subcutaneous tissue disorders) | 8 | 14
Headache (Nervous system disorders) | 11 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Gastritis (Gastrointestinal disorders) | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.